CLINICAL TRIAL: NCT07293572
Title: "The Impact of Specialized Training Course on Pre-clinical Medical Students' in Tripoli University , Performance in Disaster Medicine: A Randomized Controlled Trial"
Brief Title: "The Impact of Specialized Training Course on Pre-clinical Medical Students' in Tripoli University, Libya
Acronym: DM-Course RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tripoli (Other)
Collaborators: Libyan Red Crescent (Unknown); Faculty of Medicine - University of Tripoli (Unknown); Clinical Skills Department - Faculty of Medicine, University of Tripoli (Unknown); Medical Students' Union - Faculty of Medicine, University of Tripoli (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DM-RCT-UT-2025-Yasein-001
Record Dates: First submitted 2025-12-06; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Disaster Medicine Education and Preparedness Among Medical Students; Disaster Medicine Knowledge and Skills Training for Pre-clinical Medical Students; Disaster and Emergency Medicine Education and Preparedness Among Pre-clinical Medical Students
Keywords: medical education; pre-clinical students; RCT; training program; Libya; University of Tripoli; Tripoli; Disaster medicine; Emergency medicine
MeSH Terms: interventions — Disasters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will receive the Specialized Training Course in Disaster and Emergency Medicine (lectures + skills sessions).
  Educational Intervention → Disaster and Emergency Medicine Specialized Training Course
  Interventions: Behavioral: Specialized Training Course in Disaster and Emergency Medicine
- Control Group (No Intervention): Participants will not receive the Specialized Training Course before the post-test. They will continue their routine academic activities.

INTERVENTIONS:
Behavioral: Specialized Training Course in Disaster and Emergency Medicine — "The intervention consists of a structured Disaster and Emergency Medicine training program specifically designed for pre-clinical medical students. The program integrates theoretical modules and hands-on practical sessions delivered by university clinical skills instructors and senior members of the Libyan Red Crescent with 10-20 years of field experience. The curriculum covers disaster types, emergency response systems, first aid, psychological support, communication and coordination, outbreak prevention, volunteer safety, environmental sanitation, handling war remnants and landmines, and management of dead bodies. Training is delivered over 20-30 hours using lectures, case-based scenarios, supervised skills practice, and standardized educational materials. Learning is assessed through pre-training, mid-training, and OSCE examinations using validated scenarios reviewed by disaster medicine specialists."
  Other Names: Disaster Medicine Training Course
  Arms: Intervention Group

SUMMARY:
In recent years, Libya has faced many serious disasters that show the need for better disaster preparedness. One of the worst events was Storm Daniel in Derna in 2023, which caused heavy flooding, many deaths, and the displacement of thousands of people. Other areas, like Tarhuna and Aslitan, also suffered from floods and water leaks. These events showed that local communities are very vulnerable to natural hazards. In addition to natural disasters, Libya still faces problems from ongoing conflicts and armed clashes. These situations have caused injuries, deaths, displacement, and danger from landmines and unexploded bombs. Together, these problems show the urgent need for organized disaster medicine training, especially for medical students, who can help during emergencies. This study will test how well a structured disaster medicine training program works for pre-clinical medical students at the Faculty of Medicine, University of Tripoli. The training will include theory and practice, led by two groups: (1) university teachers who are experts in clinical skills and emergency response, and (2) the Libyan Red Crescent team, whose members have more than 10-20 years of experience in disasters and emergencies. The program will cover important topics, including: introduction to disasters, disaster response, first aid, psychological support, communication and coordination during emergencies, preventing disease outbreaks, volunteer safety, environmental sanitation, handling war remnants and landmines, and management of dead bodies. This approach will help students gain both technical skills and confidence to respond to emergencies.

The study will use a randomized controlled trial design. Students will be divided into an intervention group (receiving the training) and a control group (no training during the study). The intervention group will get at least 20-30 hours of training. To check learning, both groups will do a baseline knowledge test, then a mid-test, and an Objective Structured Clinical Examination (OSCE). The OSCE will use scenarios that were checked and approved by emergency doctors, disaster experts, and university teachers. The tests will be double-blind, meaning the students' identities will be hidden using ID codes to keep results fair. All data will be collected and analyzed following international research rules and statistical guidelines. Written consent will be obtained from all students before participating. The goal of this study is to show if structured disaster medicine training improves the knowledge, skills, and readiness of pre-clinical students. The results will help improve medical education in Libya and could also be used as a model for other countries with limited resources or ongoing conflicts, contributing to better disaster preparedness worldwide.

DETAILED DESCRIPTION:
In recent years, Libya has faced many serious disasters that show the need for better disaster preparedness. One of the worst events was Storm Daniel in Derna in 2023, which caused heavy flooding, many deaths, and the displacement of thousands of people. Other areas, like Tarhuna and Aslitan, also suffered from floods and water leaks. These events showed that local communities are very vulnerable to natural hazards. In addition to natural disasters, Libya still faces problems from ongoing conflicts and armed clashes. These situations have caused injuries, deaths, displacement, and danger from landmines and unexploded bombs. Together, these problems show the urgent need for organized disaster medicine training, especially for medical students, who can help during emergencies. This study will test how well a structured disaster medicine training program works for pre-clinical medical students at the Faculty of Medicine, University of Tripoli. The training will include theory and practice, led by two groups: (1) university teachers who are experts in clinical skills and emergency response, and (2) the Libyan Red Crescent team, whose members have more than 10-20 years of experience in disasters and emergencies. The program will cover important topics, including: introduction to disasters, disaster response, first aid, psychological support, communication and coordination during emergencies, preventing disease outbreaks, volunteer safety, environmental sanitation, handling war remnants and landmines, and management of dead bodies. This approach will help students gain both technical skills and confidence to respond to emergencies.

The study will use a randomized controlled trial design. Students will be divided into an intervention group (receiving the training) and a control group (no training during the study). The intervention group will get at least 20-30 hours of training. To check learning, both groups will do a baseline knowledge test, then a mid-test, and an Objective Structured Clinical Examination (OSCE). The OSCE will use scenarios that were checked and approved by emergency doctors, disaster experts, and university teachers. The tests will be double-blind, meaning the students' identities will be hidden using ID codes to keep results fair. All data will be collected and analyzed following international research rules and statistical guidelines. Written consent will be obtained from all students before participating. The goal of this study is to show if structured disaster medicine training improves the knowledge, skills, and readiness of pre-clinical students. The results will help improve medical education in Libya and could also be used as a model for other countries with limited resources or ongoing conflicts, contributing to better disaster preparedness worldwide.

Aims and objectives of the study :

1. To assess the baseline knowledge and preparedness of pre-clinical medical students in disaster medicine.
2. To evaluate the effectiveness of structured disaster medicine training in improving students' theoretical knowledge.
3. To evaluate the effectiveness of structured disaster medicine training in improving students' practical skills through OSCE scenarios.
4. To enhance students' confidence and readiness to participate in real-life disaster and emergency situations.
5. To provide recommendations for integrating disaster medicine training into the undergraduate medical curriculum in Libya.

any ethical issues that might arise from the proposed study and how they are be addressed :

* Voluntary participation: All students will participate voluntarily and can withdraw at any time without any penalty.
* Informed consent: Written informed consent will be obtained before any training or assessment.
* Confidentiality: Students' identities will be protected using coded IDs, and all data will be analyzed anonymously.
* Double-blinded assessments: Both intervention and control groups will be assessed under double-blind conditions to prevent bias.
* Minimizing risk: All practical exercises and OSCE scenarios will be conducted under supervision of experienced trainers from the Libyan Red Crescent, following safety guidelines.
* Compliance with international standards: The study will follow ethical guidelines and international research protocols.

ELIGIBILITY:
Inclusion Criteria:

* Pre-clinical medical students enrolled at the Faculty of Medicine, University of Tripoli.

Age between 17 and 24 years.

Able and willing to provide written informed consent.

Not previously enrolled in any formal disaster medicine or emergency medicine training course.

Available to attend all training sessions and assessment activities (pre-test, mid-test, and OSCE).

Exclusion Criteria:

* Students who have previously received structured training in disaster medicine or emergency response.

Students currently participating in another educational or training program that may influence disaster preparedness outcomes.

Students with conditions that prevent participation in simulation or OSCE activities (e.g., physical inability to perform practical tasks).

Students who refuse or are unable to provide informed consent.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in disaster medicine knowledge score | Baseline (pre-test) and immediately post-intervention.
  Assessment of participants' knowledge in disaster and emergency medicine using a validated written test covering disaster response, first aid, communication, outbreak prevention, psychological support, and safety principles. Scores from the intervention group will be compared to the control group at baseline and immediately after completion of the training. Improvement in mean score indicates higher effectiveness of the intervention.

SECONDARY OUTCOMES:
Performance in OSCE (Objective Structured Clinical Examination) | Within 1 week after completion of the training.
  Evaluation of practical disaster-response skills using standardized OSCE stations validated by emergency medicine specialists. Stations include first aid, communication, triage, psychological support, and safety procedures. Examiners are blinded to group allocation.
Self-reported disaster preparedness and confidence | Immediately after training completion.
  Student self-assessment using a structured Likert-scale questionnaire measuring perceived readiness, confidence, and ability to respond to disaster scenarios. The tool is adapted from previously validated disaster preparedness surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Elhadi, MD, Principal Investigator — Faculty of Medicine - University of Tripoli
Locations (1):
- Faculty of Medicine, University of Tripoli, Tripoli, Libya

IPD SHARING:
Plan to Share IPD: No
The study involves educational assessments of pre-clinical medical students, including knowledge tests and OSCE performance. The data are sensitive and linked to individual participants. Therefore, individual participant data (IPD) will not be shared with other researchers to protect student privacy.